CLINICAL TRIAL: NCT07359833
Title: Effects of FiO2 Adjustment on Hyperoxia Biomarkers and Postoperative Complications Using Oxygen Reserve Index During One-lung Ventilation
Brief Title: Oxygen Reserve Index Guided FiO₂ Titration in One-Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Bugra AYKENAR, Anesthesia resident, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziU-AR-BA-01
Record Dates: First submitted 2026-01-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2022-08

CONDITIONS: One Lung Ventilation in Thoracic Surgery
Keywords: One-Lung Ventilation; oxygen reserve index; Hyperoxia; Thoracic surgery; Oxidative stress; Oxygen
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel-group clinical trial comparing ORi-guided intraoperative FiO₂ titration with conventional oxygen management in adult patients undergoing thoracic surgery with one-lung ventilation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ORi group. (Experimental): In this group, intraoperative FiO₂ was titrated according to predefined Oxygen Reserve Index (ORi) thresholds during one-lung ventilation and all intraoperative period, with the aim of maintaining adequate oxygenation while avoiding unnecessary hyperoxia.
  Interventions: Device: Oxygen Reserve Index (ORi)-guided oxygen titration
- Non-ORi group (No Intervention): In this group, intraoperative FiO₂ was adjusted based solely on pulse oximetry (SpO₂) monitoring, without the use of Oxygen Reserve Index (ORi) guidance.

INTERVENTIONS:
Device: Oxygen Reserve Index (ORi)-guided oxygen titration — FiO₂ adjusted intraoperatively according to predefined ORi thresholds during thoracic surgery and one lung ventilation period.
  Arms: ORi group.

SUMMARY:
One-lung ventilation (OLV) is routinely used during thoracic surgery to facilitate surgical exposure but is associated with an increased risk of intraoperative hypoxemia. To prevent hypoxia, high fractions of inspired oxygen (FiO₂) are commonly administered; however, excessive oxygen delivery may lead to hyperoxia and oxidative tissue injury. The Oxygen Reserve Index (ORi) is a novel, noninvasive monitoring parameter that provides real-time information on moderate hyperoxia and may allow more precise titration of FiO₂ during anesthesia.

The aim of this prospective, randomized clinical trial is to evaluate whether ORi-guided intraoperative oxygen management can reduce oxygen exposure during OLV without increasing hypoxemia and to assess its effects on oxidative stress biomarkers and postoperative outcomes. Adult patients undergoing elective thoracic surgery with OLV are randomized to receive either ORi-guided FiO₂ titration or conventional oxygen management. Oxidative stress biomarkers and postoperative pulmonary complications are compared between groups.

DETAILED DESCRIPTION:
One-lung ventilation is an essential component of thoracic anesthesia but poses significant challenges in maintaining adequate oxygenation. In clinical practice, high FiO₂ levels are often applied to prevent hypoxemia; however, prolonged exposure to hyperoxia has been associated with increased oxidative stress, inflammatory responses, and potential tissue damage. Despite growing awareness of oxygen toxicity, optimal intraoperative oxygen titration strategies during OLV remain poorly defined.

The Oxygen Reserve Index is derived from multiwavelength pulse oximetry and provides continuous, noninvasive information on moderate hyperoxia (corresponding to arterial oxygen tensions above normoxia but below severe hyperoxia). ORi monitoring may enable anesthesiologists to titrate FiO₂ more precisely, thereby avoiding unnecessary oxygen exposure while maintaining adequate oxygenation.

In this prospective, randomized clinical trial, adult patients scheduled for elective thoracic surgery requiring OLV are allocated to either an ORi-monitored group or a control group. In the ORi group, FiO₂ is adjusted intraoperatively according to predefined ORi thresholds, whereas in the control group FiO₂ is managed according to standard clinical practice based on pulse oximetry. Blood and tracheal aspirate samples are collected preoperatively and at predefined postoperative time points to measure interleukin-6, superoxide dismutase, and malondialdehyde levels as markers of inflammation and oxidative stress. Postoperative pulmonary complications and surgical site infections are recorded during intensive care unit and ward follow-up.

This study aims to determine whether ORi-guided oxygen titration during OLV can safely reduce intraoperative oxygen exposure and to clarify its impact on biochemical markers of oxidative stress and clinical outcomes such as postoperative pulmonary complications and surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18-85 years Elective case Thoracic surgeries performed with one-lung ventilation using a double-lumen endotracheal tube Left ventricule ejection fraction(LVEF)>45%

Exclusion Criteria:

* heart failure (LVEF) < 45% severe valvular disease admission as an emergency case history of prior lung resection presence of peripheral arterial disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Mean intraoperative FiO₂ | From anesthesia induction to the extubation
  The primary outcome is the mean fraction of inspired oxygen (FiO₂) administered during one-lung ventilation and throughout the entire duration of surgery, recorded continuously intraoperatively and compared between the ORi-guided and conventional oxygen management groups.

SECONDARY OUTCOMES:
Oxidative stress biomarkers (IL-6, SOD, MDA) | Anesthesia induction, extubation, postoperative 12th hour, postoperative 24th hour
  Changes in serum and tracheal aspirate levels of interleukin-6, superoxide dismutase, and malondialdehyde assessed at four time points. Serum biomarker levels are measured at anesthesia induction and at the 12th and 24th postoperative hours, while tracheal aspirate biomarker levels are measured at extubation. Results are compared between the ORi and Non-ORİ groups.
Postoperative pulmonary complications | up to 2 weeks
  Incidence of postoperative pulmonary complications, including prolonged drainage, hemothorax, bronchopleural fistula, reintubation, atelectasis, bronchopneumonia, and acute respiratory distress syndrome, assessed during intensive care unit and ward follow-up.
Surgical site infections | up to 2 weeks
  Incidence of surgical site infections recorded during postoperative hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Buğra Aykenar, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data generated during this study may be made available for use in future meta-analyses upon reasonable request to the corresponding author.

REFERENCES:
- [Result] Saracoglu A, Yamansavci Sirzai E, Yildizeli B, Yuksel M, Aykac ZZ. Oxygen reserve index guided oxygen titration in one lung ventilation with low fresh gas flow. Turk J Med Sci. 2021 Oct 21;51(5):2413-2419. doi: 10.3906/sag-2009-149. PMID 34051711